CLINICAL TRIAL: NCT00070785
Title: Comprehensive Epitope Mapping of the Epstein-Barr Virus Latent Membrane Protein-2 in Ethnically Diverse Populations
Brief Title: Protein Studies of the Epstein-Barr Virus in Ethnically Diverse Populations
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040007; 04-CC-0007; NCT00897156 (obsolete NCT alias)
Record Dates: First submitted 2003-10-07; First posted 2003-10-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-04-21

CONDITIONS: Epstein-Barr Virus Infections
Keywords: Nasopharyngeal Cancer; EBV Virus; Epitope Mapping; Epstein-Barr Virus; Latent Protein-2; Healthy Volunteer; HV
MeSH Terms: conditions — Epstein-Barr Virus Infections; Nasopharyngeal Neoplasms

SUMMARY:
This study will evaluate the ability of people of different ethnic backgrounds to develop immune responses against the Epstein-Barr virus (EBV). A common virus, EBV is present in 90 percent of healthy people and usually does not cause problems. Most people are infected in childhood, have no symptoms, and are unaware of their infection. People infected as adolescents or adults may develop infectious mononucleosis, which usually resolves completely. However, in immune suppressed people, like those who have had a transplant, EBV can cause fatal cancers. It can also cause certain cancers such as Burkitt's lymphoma, Hodgkin's lymphoma, and nasopharyngeal carcinoma in people who are not immune suppressed. Nasopharyngeal carcinoma is 100 times more common in people of Asian origin (particularly southern Chinese) compared with Caucasians. This difference may be the result of genetic, rather than environmental, factors. This study will examine whether the same proteins produced by EBV in the cancer cells react differently in people of different ethnic background in a way that could explain the differences in predisposition for this disease.

Healthy normal volunteers 18 years of age and older of Caucasian or Chinese ancestry may be eligible for this study. Candidates of Chinese ancestry must be born in China (including Taiwan, Hong Kong, and Singapore, or be first generation offspring of parents born in these places).

Participants will have a blood sample drawn and will undergo lymphapheresis - a procedure for collecting large numbers of white blood cells called lymphocytes. The blood sample is tested for blood counts and HLA type, a genetic marker of the immune system. HLA molecules help determine the way the body's immune cells respond to virus. HLA typing is similar to blood typing. Usually done to match stem cell or organ transplants, HLA testing may also be used to try to identify factors associated with an increased risk of certain diseases or conditions. HLA type is strongly associated with ethnic background.

For lymphapheresis, blood is collected through a needle in an arm vein, similar to donating blood. The blood flows from the vein through a catheter (plastic tube) into a machine that separates it into its components by centrifugation (spinning). The white cells are removed and the rest of the blood (red cells, plasma and platelets) is returned to the body through a needle in the other arm. The procedure takes 2 to 3 hours. The collected white cells are used for research for this study, including the ability to react to EBV proteins, and are then destroyed.

DETAILED DESCRIPTION:
Epstein Barr virus (EBV) can induce in immune compromised patients fatal lymphoproliferative lesions that regress upon reversion of immune suppression or adoptive transfer of EBV-specific CD8+ T cells. EBV can also induce neoplastic lesions in immune competent hosts including Burkitt's lymphoma, Hodgkin's disease and nasopharyngeal cancer (NPC). EBV-specific CD8+ T cell responses can occur in patients with these cancers that are qualitatively similar but quantitatively diminished compared to EBV-primed normal individuals. Although these cancers share several features, they are characterized by divergent patterns of expression of EBV proteins. In particular, NPC expresses preferentially the latent membrane protein (LMP) 2 with or without expression of LMP 1 and intermediate expression of the Epstein-Barr nuclear antigen. Thus, there is interest to develop LMP 2-directed immunizations for patients with NPC with the hope that enhancement of the insufficient natural immunity may lead to tumor regression. Since, the incidence of NPC is tightly associated with ethnic background (principally Southern Chinese) and Human Leukocyte Antigen (HLA) phenotype, diverse populations may display distinct reactivity patterns toward EBV epitopes that may in turn be responsible for their respective predisposition to acquire NPC. Although, several LMP 2 epitopes have been described, to our knowledge, no systematic mapping across diverse ethnicity complemented with high-resolution HLA typing has ever been done. We, therefore, propose to map immune dominant epitopes of LMP 2 in EBV primed normal individuals of Caucasian or Asian (Chinese) ethnicity by measuring interferon (IFN)-gamma transcript levels in circulating lymphocytes exposed to a library of overlapping nonamer peptides encompassing the full sequence of LMP 2. High resolution, sequence-based HLA typing will complement the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Normal volunteers, age greater than or equal to 18 years of Caucasian or Chinese ancestry will be eligible for the study. Chinese ancestry will be defined as being born in China (including Taiwan, Hong Kong and Singapore) or being first generation offspring of parents born in China (including Taiwan, Hong Kong and Singapore).

ECOG performance status of 0 or 1.

Individuals must weigh at least 110 pounds.

Potential participants must pass the criteria for blood donors established by the American Association of Blood Banks according to the routine screening performed within the Department of Transfusion Medicine.

Potential participants should pass a brief physical exam to exclude potential cardiac problems.

WBC 3000/mm(3) or greater.

Platelet count 90,000 mm(3) or greater.

Negative pregnancy test

Ante-cubital veins compatible with the apheresis process. Apheresis center nurses will assess the ante-cubital veins of all subjects prior to enrollment. If their veins are judged to be too small to support the intravenous catheter required for the procedure, they will be excluded. If at the time of each apheresis procedure the nurses are unable to obtain adequate ante-cubital vein access, the subject will be excluded.

Evidence of previous exposure to EBV infection will not represent inclusion criteria.

EXCLUSION CRITERIA:

Potential participants will be excluded:

Who are undergoing or have undergone in the past 3 weeks any form of systemic therapy that may affect immune function.

Who have active systemic infections, autoimmune disease or any known immunodeficiency disease.

Who require systemic steroid therapy.

Who are pregnant.

Who are positive for hepatitis B (s)AG or HIV antibody (because of possible immune effects of these conditions). HIV testing will be performed prior to enrollment.

Who have any form of active primary or secondary immune deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-10-06; Study Completion 2008-04-21

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Heslop HE, Rooney CM. Adoptive cellular immunotherapy for EBV lymphoproliferative disease. Immunol Rev. 1997 Jun;157:217-22. doi: 10.1111/j.1600-065x.1997.tb00984.x. PMID 9255632